CLINICAL TRIAL: NCT00283010
Title: Improvement in Memory With Plasticity-Based Adaptive Cognitive Training (IMPACT)
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: Mayo Clinic (Other); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OUT-105-2005
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Aging
Keywords: cognitive enhancement; memory; auditory memory; speech; computerized; cognitive decline
MeSH Terms: conditions — Speech; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Experimental Treatment (Experimental): Computerized Plasticity-Based Adaptive Cognitive Training
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training
- Active Control (Active Comparator): Educational DVDs
  Interventions: Other: Educational DVDs

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training
  Other Names: BrainHQ; Brain Fitness Program
  Arms: Experimental Treatment
Other: Educational DVDs
  Arms: Active Control

SUMMARY:
The primary objective of this study is to evaluate the effects of a computer-based training program on the memory and cognitive abilities of mature individuals undergoing healthy aging.

DETAILED DESCRIPTION:
The computer-based training program is focused on speech reception to strengthen an individual's memory for speech. This type of training program was chosen because speech perception and memory are crucial elements of human communication and losses in this area are often the first signal of overall cognitive decline.

Subjects meeting eligibility criteria and providing written, informed consent are randomized to one of two 40-session, computerized training programs.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older at the time of consent.
* Mini-Mental State Examination (MMSE) score of 26 or higher.
* Fluent English speaker. For the purposes of this study, fluency will be defined as living in an English speaking country and attending an English speaking school by the age of six (participants will demonstrate fluency by reading aloud a selected paragraph).
* Visual capacity adequate to read 14 point type (participants will demonstrate visual capacity by reading aloud a selected sentence).
* Adequate hearing capacity. (Participants will demonstrate by repeating a series of words spoken by the screening clinician; the words will be spoken while a view of the clinician's mouth is obstructed to prevent lip-reading.)
* Willing and able to commit to the 6-month time requirement of the entire study period with an emphasis on availability for the 8-10 week computer based training.

Exclusion Criteria:

* Mini-Mental State Examination (MMSE) score of 25 or lower.
* Self-report of current diagnosis or history of major neurological illness. Specifically:

  * Alzheimer's disease
  * Parkinson's disease
  * Multiple sclerosis
  * Amyotrophic lateral sclerosis
* Self-report of current diagnosis or history of psychiatric illness. Specifically:

  * Major depressive disorder
  * Bipolar disorder
  * Schizophrenia
  * Post traumatic stress disorder
  * Obsessive-compulsive disorder
* Self-reported history of psychiatric hospitalization.
* History of a stroke, transient ischemic attack (TIA), or traumatic brain injury within the past year; or lifetime history of stroke, TIA, or traumatic brain injury that has left residual expressive or receptive language problems. Traumatic brain injuries include, but are not limited to: concussion with loss of consciousness; head trauma with loss of consciousness; persistent migraines (persistent being defined as a predictable pattern occurring more frequently than every other month); and history of seizure disorder.
* Fibromyalgia or symptoms of tremor severe enough to prevent the use of a computer mouse or other pointing device. Clinician to observe participant during signature of consent form, during drawing portion of Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) assessment, and to directly ask participant as instructed in the Body Image Ideals Questionnaire (BIQ) to make tremor assessment.
* Self-report of current substance abuse, including alcoholism.
* Current use, or use within the past 3 months, of medications with substantial central nervous system (CNS) effects, including acetylcholinesterase inhibitors and medications with either anticholinergic or antidepressant properties.
* Behaviors during screening or baseline visits that, in the judgment of the screening clinician, are likely to present significant problems for the trainers in the in home setting may be excluded at the discretion of the clinician. Such behaviors include significant uncooperative behavior, significant rudeness or temper management problems, or inappropriate physical conduct.
* Unable to perform neuropsychological evaluations.
* Participant is not capable of giving informed consent or is unable to comprehend and/or follow instructions.
* Participant is enrolled in a concurrent clinical study that could affect the outcome of this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 487 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Cognitive effects of training | 6 months

SECONDARY OUTCOMES:
Safety effects of computer-based training | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Henry W Mahncke, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- Posit Science Corporation, San Francisco, California, United States

REFERENCES:
- [Result] Smith GE, Housen P, Yaffe K, Ruff R, Kennison RF, Mahncke HW, Zelinski EM. A cognitive training program based on principles of brain plasticity: results from the Improvement in Memory with Plasticity-based Adaptive Cognitive Training (IMPACT) study. J Am Geriatr Soc. 2009 Apr;57(4):594-603. doi: 10.1111/j.1532-5415.2008.02167.x. Epub 2009 Feb 9. PMID 19220558
- [Result] Zelinski EM, Spina LM, Yaffe K, Ruff R, Kennison RF, Mahncke HW, Smith GE. Improvement in memory with plasticity-based adaptive cognitive training: results of the 3-month follow-up. J Am Geriatr Soc. 2011 Feb;59(2):258-65. doi: 10.1111/j.1532-5415.2010.03277.x. PMID 21314646
- [Result] Zelinski EM, Peters KD, Hindin S, Petway KT 2nd, Kennison RF. Evaluating the relationship between change in performance on training tasks and on untrained outcomes. Front Hum Neurosci. 2014 Aug 13;8:617. doi: 10.3389/fnhum.2014.00617. eCollection 2014. PMID 25165440